CLINICAL TRIAL: NCT05161065
Title: Comparison of QT Interval Readings Between Smartwatch Combined With Cardiologs Artificial Intelligence and 12-lead ECG in Subjects Hospitalized for Antiarrhythmic Drug Initiation and Follow-up
Brief Title: Comparison of QT Interval Readings Between Smartwatch Combined With Cardiologs Artificial Intelligence and 12-lead ECG
Status: Completed | Type: Observational
Sponsor: Cardiologs Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: WatchQT
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Cardiologs — Apple Watch recordings interpreted by Cardiologs AI done simultaneously with each 12-lead ECG
  Other Names: Apple Watch

SUMMARY:
The WatchQT study will compare the performance of a smartwatch combined with Cardiologs ECG AI Analysis system in monitoring corrected QT (QTc) intervals with that measured on a manually read 12-lead ECG in subjects with Normal Sinus Rhythm (NSR) during antiarrhythmic drug (AAD) initiation and follow-up at the hospital.

DETAILED DESCRIPTION:
The WatchQT Study is a prospective, non-significant risk, non-randomized, monocentric, open, comparative, concordance pilot study.

Under subject consent, subjects hospitalized for AAD initiation and monitoring will have smartwatch ECG recordings done simultaneously with 12-lead ECG measurements before and after drug administration twice a day, in accordance with the existing in-stay subject monitoring protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over 22, able and willing to participate in the study
2. Subjects who are admitted to the hospital in NSR or AF and are eligible for AAD (class Ia or class III) dose initiation or re-initiation.
3. Subjects having read the patient information letter and provided his/her consent to participate in writing, by dating and signing the informed consent prior to any trial-related procedure being conducted

Exclusion Criteria:

1. Subjects with Cardiac Implantable Electronic Devices (CIED)
2. Pregnant or breast-feeding subjects

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 to 50 Subjects: Subjects who are being hospitalized for antiarrhythmic drug (AAD) initiation and monitoring per standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Concordance between QTc intervals (in ms) measured by smartwatch combined with Cardiologs AI and that measured by manually read 12-lead ECG | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Concordance between QTc intervals measured by smartwatch combined with Cardiologs AI and that measured by manually read 12-lead ECG for each measurement done during NSR. The Bazett (QTcB in ms) and Fridericia (QTcF in ms) methods will be used to correct QT intervals

SECONDARY OUTCOMES:
Description of the sensitivity and specificity of the smartwatch combined with Cardiologs AI | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Description of the sensitivity and specificity of the smartwatch combined with Cardiologs AI in determining subjects at risk of AAD induced ventricular arrhythmia compared to that identified by manually read 12-lead ECG in subjects with a prolonged QTc > 500 ms and/or subjects with a QTc prolongation of > 15% after their initial AAD dose
Concordance between QTcB and QTcF intervals measured by the different methods | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Concordance between QTcB and QTcF intervals measured by the different methods (smartwatch combined with Cardiologs AI, smartwatch read manually, 12-lead read manually, lead 1 from 12-lead read manually and automated interpretation of the 12 lead ECG machine)
Description of the QTc interval measurements in NSR | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Description of the QTc interval measurements in NSR as a function of timepoints by the different methods
Quantitative analysis to determine the interobserver variability | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Quantitative analysis to determine the interobserver variability in QTc interval measurements by the smartwatch and 12-lead ECG manual readings
Description of the QT interval defined as uncertain by the smartwatch combined with Cardiologs AI | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Description of the QT interval defined as uncertain by the smartwatch combined with Cardiologs AI
Descriptive analysis of QT interval measurements in AF measured by smartwatch combined with Cardiologs AI and manually read 12-lead ECG | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  .Descriptive analysis of QT interval measurements in AF measured by smartwatch combined with Cardiologs AI and manually read 12-lead ECG at each timepoint and overall.
Analysis of QT interval measured in subsets of subjects with and without wide QRS | Readings taken simultaneously right before and 2-3 hours after drug administration during hospitalization
  Patient with wide QRS is determined as a QRS>120ms at D0 from automated interpretation of the 12-lead ECG machine. The analysis will be done in subset of 2 groups according to the QRS measured as wide or not machine

CONTACTS AND LOCATIONS:
Overall Officials: Jagmeet Singh, MD ScM DPhil, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No